CLINICAL TRIAL: NCT00628784
Title: Endoesophageal Cryotherapy: A New Technique For Ablating Barrett's Esophagus And Early Stage Esophageal Cancer
Brief Title: Endoesophageal Cryotherapy For Ablating Barrett's Esophagus and Early Stage Esophageal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: CSA Medical, Inc. (Industry)
Responsible Party: LTC John David Horwhat MD FACG, Gastroenterology Service Walter Reed Army Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-14034
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Barrett's Esophagus
Keywords: Dysplasia; Ablation; Squamous dysplasia; Early esophageal adenocarcinoma; Cryotherapy
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Specialized intestinal metaplasia (Barrett's esophagus) documented via endoscopic esophageal biopsy, with standard surveillance biopsies (four-quadrant biopsies obtained every 2-cm the entire length of the specialized intestinal metaplasia in the esophagus) performed within the past two years prior to study enrollment. Biopsies show either low grade dysplasia, indeterminate for dysplasia, or no dysplasia.
  Interventions: Procedure: Endoscopic spray cryotherapy
- Group 2 (Experimental): Diagnosis of Barrett's esophagus and high grade dysplasia or intramucosal carcinoma. Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney, or liver disease; or refusal of surgical intervention. CT scan demonstrating no evidence of advanced esophageal cancer (extension into or through the wall or lymph node involvement). Endoscopic ultrasound* (EUS) demonstrating no evidence of metastatic lymph node involvement or extension of carcinoma beyond the mucosa (T1).
  Interventions: Procedure: Endoscopic spray cryotherapy
- Group 3 (Experimental): Diagnosis of esophageal carcinoma (T1smN0 or T2N0 via EUS). Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney, or liver disease; or refusal of surgical intervention. CT scan demonstrating no evidence of advanced esophageal cancer (extension into or through the wall or lymph node involvement).
  Interventions: Procedure: Endoscopic spray cryotherapy
- Group 4 (Experimental): Diagnosis of severe dysplasia within esophageal squamous mucosa on pathology review. Deemed inoperable based on the following criteria: co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention. CT scan demonstrating no evidence of advanced esophageal cancer (extension into or through the wall or lymph node involvement). EUS with no evidence of metastatic lymph node involvement or extension of carcinoma beyond the mucosa.
  Interventions: Procedure: Endoscopic spray cryotherapy

INTERVENTIONS:
Procedure: Endoscopic spray cryotherapy — A special orogastric venting tube is passed alongside the endoscope and the cryocatheter then used to perform cryotherapy. Liquid nitrogen is sprayed through the catheter to achieve a uniform white frost in a hemicircumferential sector for 10 seconds. A thaw time of 45-60seconds is observed. This freeze-thaw cycle is repeated x 3 for a total of 40sec cryotherapy per segment. This therapy is repeated every 6 weeks until visible re-epithelialization is seen or a maximum of 6 sessions. Once a squamous lining is seen, biopsies are taken throughout the original area to assess for buried Barretts. If none is seen, followup with 4 quadrant q2cm biopsies are taken at 3,6,9,12, 18, 24, 36, 48 months.
  Other Names: Cryotherapy
  Arms: Group 1; Group 2; Group 4
Procedure: Endoscopic spray cryotherapy — After passing a special orogastric venting tube, the cryocatheter is used to spray liquid nitrogen onto the tumor to achieve a white frost (frozen state) for 20 seconds. A 45-60 sec thaw is allowed and then retreatment x 2 for a total of 60 seconds therapy per session. Repeat treatments are permitted every 2 weeks for a maximum of 8 treatments.
  Other Names: Cryotherapy
  Arms: Group 3

SUMMARY:
In this prospective single center study, up to 25 patients with Barrett's esophagus with LGD or no dysplasia (Group 1), 25 patients with HGD/IMCA (Group 2), 25 patients with esophageal carcinoma confined to the esophageal wall (Group 3) and 25 patients with severe esophageal squamous dysplasia (Group 4) will be treated with endoscopic cryotherapy. This study is single arm and no blinding will be utilized. Interim analysis of the data will be reviewed with a DCI statistician after 14 patients in each group have been treated with cryotherapy and if safety and efficacy is documented to that point in time, we will request the ability to extend the enrollment to a maximum allowable amount of 25 patients per group. The proposed study duration is seven years, allowing two years for patient enrollment and 5 years for post treatment follow-up. Study duration per patient will total approximately six years.

Patients with Barrett's esophagus with no dysplasia or low grade dysplasia (group 1) will be treated with cryotherapy at six week intervals until Barrett's mucosa is ablated or six treatments are administered. Patients with Barrett's HGD and IMCA or severe esophageal squamous dysplasia (groups 2 and 4) will be treated with cryotherapy at six-week intervals until Barrett's mucosa is ablated or six treatments are administered. More advanced mass lesions are typically more difficult to eradicate with ablative therapies and may progress faster than patients with IMCA, therefore, patients with more advanced cancer (group 3) will be treated every 2 weeks until the lesion is eradicated up to eight treatments.

After cryotherapy treatment is complete (i.e. the esophagus has re-epithelialized with normal squamous epithelium for Groups 1, 2, 4 and the tumor is locally controlled/absent in Group 3), patients will be assessed by endoscopy and biopsy every three months for one year, every six months for two years, then annually for two years (flow sheet - appendix 1; study schedule - appendix 2).

DETAILED DESCRIPTION:
Baseline evaluation will include the following ( all are considered standard of care except # 8 ):

1. Informed consent.
2. Evaluation of inclusion/exclusion criteria
3. Demographics- date of birth, age, gender, ethnicity
4. Medical history and physical exam
5. Imaging (groups 2, 3 and 4) i. CT scan of the chest and abdomen with oral and intravenous contrast (if not allergic) ii. Endoscopic Ultrasound, with evaluation of the esophageal wall and mediastinum and upper abdomen for evidence of abnormal lymph nodes. Suspicious lymph nodes (round, hypoechoic, homogeneous, > 5mm) will undergo EUS-guided fine needle aspiration if appropriate, as deemed by the principal investigator.
6. Pathology review (groups 2 and 4) - two independent reviewers, including at least one from the WRAMC Pathology Department, will review the pathology slides from esophageal biopsies. This review will serve to confirm the diagnosis of Barrett's esophagus with high grade dysplasia and/or IMCA for agreement of the diagnosis of adenocarcinoma and the degree of dysplasia.
7. Presentation at Tumor Board prior to entering the protocol (groups 2, 3 and 4).
8. Dysphagia score (see Appendix 4) is for research purposes.

Prior to cryotherapy:

As part of the research protocol, all patients will be treated with high dose proton pump inhibitor (PPI) (lansoprazole 30mg, esomeprazole 40mg, pantoprazole 40mg, omeprazole 40mg or rabeprazole 40mg) BID for maximal acid suppression until complete ablation is achieved or the patient exits the study. All of these agents are considered equally effective at the doses listed with no one agent considered superior. Treatment with these research doses will begin at least one week prior to the first cryotherapy session. Pre-enrollment standard doses of PPI will be restarted once the patient enters the surveillance phase or exits the study. Care will be taken to avoid, if possible, any potentially toxic medications to the esophageal mucosa (i.e. non-steroidal anti-inflammatory drugs, bisphosphonates, potassium supplements).

EGD/Cryotherapy Patients will be scheduled for EGD with cryotherapy on designated days when support for the cryotherapy device is available according to the study timeline (Appendix 2). A commitment from the CSA Medical Inc. (Baltimore, MD) will provide technical support for sessions to allow patients timely treatment.

Patients will prepare for EGD in the standard fashion using an overnight fast with only sips of clear liquids and required medications allowed up to 2 hours before the procedure. Patients will be interviewed prior to the procedure using a standardized questionnaire (Appendix 3). This questionnaire will assess overall sense of well-being, general state of health, ability to perform activities of daily living, and ability to eat. It will specifically solicit symptoms of chest pain, irregular heart rate, shortness of breath, dysphagia or odynophagia. A dysphagia score will also be measured (appendix 4).

Moderate sedation with intravenous meperidine or fentanyl and midazolam will be administered and staff investigators will perform the EGD using a therapeutic upper endoscope with adherence to standard protocol. A 14 to 18 French nasogastric tube which has been modified with decompression ports spanning the distal 12 inches of the tube (to allow decompression of both the stomach and the esophagus) will be placed into the stomach under direct visualization. This is connected to continuous suction to allow decompression during the cryotherapy procedure. During the procedure an assistant will monitor and record the heart rate, blood pressure and oxygen saturation per WRAMC moderate sedation guidelines.

All subjects will be treated with narcotic analgesics and anti-emetics as needed after each procedure.

Groups 1, 2 and 4 At the first procedure, the most proximal edge of the squamocolumnar junction (SCJ) and the tips of the gastric folds (gastroesophageal junction of GEJ) will be marked with a submucosal tattoo of India ink (SPOT, GI Supply, Camp Hill, PA) using a standard sclerotherapy needle (if not already performed). The ink tattoo will guide measurement of response to ablation and sampling the neo-squamous segment for residual Barrett's during follow up exams. For severe esophageal squamous dysplasia, the tattoo will be applied at the proximal and distal margins of the dysplastic area. If not allergic to iodine, Lugol's solution will be used to stain the squamous mucosa during the exam to outline the area of severe squamous dysplasia and guide the tattoo placement. Lugol's is chosen since normal squamous, but not dysplasia or carcinoma stains with this vital stain. These marks are placed for research purposes only and help to ensure that accurate measurements to assess the change of Barrett's segment with therapy are recorded. (30) The location of the squamocolumnar junction (SCJ), the esophagogastric junction (EGJ) and diaphragmatic hiatus (DH) will be documented in terms of centimeters from the incisors. Any islands of squamous tissue within the Barrett's segment will be photographed, measured, and recorded. If the SCJ is not well visualized, chromoendoscopy with Lugol's solution, which highlights the squamous epithelium, will be performed.

The cryocatheter is passed into the therapeutic channel of the endoscope and extended one cm beyond the distal tip of the scope. Liquid nitrogen is sprayed through the cryocatheter, which causes a white frost (cryoburn) on the adjacent mucosa. The most distal aspect of the Barrett's esophagus segment is treated first and the endoscope is slowly withdrawn proximally, maneuvering the tip of the cryocatheter such that the cryoburn is extended to "paint" a white frost cryoburn circumferentially. The spray will be applied for duration of 10 seconds as measured by the integrated device timer. During each cryotherapy session, the process will be repeated up to four times in piecemeal fashion such that for any given area treated it will be maintained in a frozen state for a total of 40 seconds. A frozen state will be defined as mucosa appearing white.

At the completion of the endoscopic procedure, the patients are monitored in our recovery area until completely awake, alert and able to be discharged according to our standard conscious sedation policy. Following discharge from the endoscopy suite, patients will be contacted in one week by telephone to assess for any immediate complications. A questionnaire will be completed by the study physician or nurse (appendix 3). Patients will be seen the same day in the clinic or endoscopy center for any serious concerns (patient or study personnel).

Patients will return in 6 weeks (groups 1, 2 and 4) for reassessment with a repeat EGD and cryotherapy for residual Barrett's mucosa. The interview questionnaire and dysphagia score will be repeated before each EGD. The location of the SCJ, the EGJ and DH and dysplastic region will be recorded and photographed to characterize the precise size and location of any islands of squamous tissue within the Barrett's segment. If there is gross evidence of mucosal injury due to the previous cryotherapy (any mucosal break including erosions, tears, or ulcers) the procedure will be terminated and further ablation will be held for an additional 2 weeks. If there is no gross evidence of esophageal mucosal injury, cryotherapy will be repeated. The process will continue until complete ablation of the Barrett's mucosa has been achieved or the maximum number of treatment sessions has been performed (8 treatments total).

When it appears endoscopically that all or nearly all of the mucosa has been replaced with normal appearing squamous mucosa, a biopsy or several biopsies may be taken at the discretion of the endoscopist of any suspicious areas to confirm that cryotherapy has been completed. When such "quick look" biopsies have been taken, no cryotherapy will be performed that day.

If the pathology results return revealing sub-squamous intestinal metaplasia or dysplasia, cryotherapy may be resumed two weeks after the biopsies had been taken (to allow adequate time for the mucosa to have healed). If the biopsy confirms resolution, the patient will then be scheduled for post-cryotherapy surveillance.

Biopsies taken during these endoscopies will be used only for the clinical purpose of assessing the patient's histologic response to cryotherapy. As such, no excess tissue will be collected or stored for any purposes.

Group 3:

Group 3 patients will undergo cryotherapy with intent to ablate the neoplasia. Group 3 patients with long segment Barrett's esophagus will undergo ablation of only the nodular areas and/or mass lesions. Flat Barrett's will not be treated. The mass lesion will be treated in its entirety until frozen or up to 20 seconds. This will be repeated for a total treatment time of 60 seconds.

Follow up endoscopy to allow repeat treatment with cryotherapy will be every two weeks until the lesion is eradicated or is treated up to 8 times, whichever comes first. These patients are being offered more aggressive therapy (every 2 weeks rather than every 6 weeks), due to the presence of more advanced disease. Treatment will be withheld for evidence of active ulceration and will not be resumed until this has healed. When it appears endoscopically that the cancer has been eradicated and all or nearly all of the mucosa has been replaced with normal appearing squamous mucosa, a biopsy or several biopsies may be taken at the discretion of the endoscopist of any suspicious areas to confirm that cryotherapy has been completed. When such "quick look" biopsies have been taken, no cryotherapy will be performed that day. If the pathology results return revealing sub-squamous intestinal metaplasia, dysplasia or cancer, cryotherapy may be resumed. If the biopsy confirms resolution, the patient will then be scheduled for post-cryotherapy surveillance.

Biopsies taken during these endoscopies will be used only for the clinical purpose of assessing the patient's histologic response to cryotherapy. As such, no excess tissue will be collected or stored for any purposes. No blood will be drawn for this study.

The initial EGD procedures are estimated to require up to 45 minutes to perform due to the possible need to perform Lugol's staining and/or India ink marking of the esophagus. Subsequent re-treatment EGD's are estimated to require no more than 30 minutes to perform. An EGD that reveals healing where only "quick look" biopsies are taken will take no more than 10 minutes to perform.

ELIGIBILITY:
Inclusion Criteria:

* ** You must be eligible for care within the Department of Defense (DEERS eligible) to be enrolled into this protocol **
* Per Groups 1,2,3,4 (above)
* Specifically:
* Diagnosis of specialized intestinal metaplasia (Barrett's esophagus) with either low grade, indeterminate or no dysplasia (Group 1)
* high grade or intramucosal cancer and deemed inoperable based on co-morbid conditions such as severe heart, lung, kidney or liver disease; or refusal of surgical intervention; CT scan and EUS demonstrating no evidence of trans-mural tumor or lymph node involvement; pathology review of esophageal biopsies by 2 independent reviewers to include 1 from the Walter Reed Army Medical Center Pathology Department; presentation at tumor board (Group 2)
* T1smN0 or T2NO adenocarcinoma arising in Barrett's esophagus and all criteria as for group 2 (Group 3)
* diagnosis of severe squamous dysplasia and all criteria as for group 2 (Group 4)

Exclusion Criteria:

* Not eligible for care within the Department of Defense medical system
* Age less than 18 years or greater then 85 years (at time of entry)
* Co-morbid illness expected to cause death within 6 months
* Pregnancy (as determined by urine HCG)
* Medically unfit or other contraindications to tolerate upper endoscopy
* Inability to tolerate therapy with a proton pump inhibitor
* Refusal or inability to give consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Confirm the feasibility and safety of endoscopic cryotherapy in patients with Barrett's esophagus with LGD, HGD, intramucosal cancer and in patients with severe squamous dysplasia. | These outcomes are measured at each endoscopy, with limits set on the number of procedures that can be done based on group assignment.

SECONDARY OUTCOMES:
Assess the incidence of side effects, complications, adverse events and number of treatment sessions needed to reach primary endpoints. | Measured throughout the protocol during the treatment phase with cryotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: John D Horwhat, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States